CLINICAL TRIAL: NCT01335932
Title: A Randomized Double-Blind Placebo-Controlled Trial of Ganciclovir/Valganciclovir for Prevention of Cytomegalovirus Reactivation in Acute Injury of the Lung and Respiratory Failure (The GRAIL Study)
Brief Title: Ganciclovir/Valganciclovir for Prevention of CMV Reactivation in Acute Injury of the Lung and Respiratory Failure
Acronym: GRAIL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Boeckh, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 7217; U01HL102547 (NIH)
Record Dates: First submitted 2011-04-13; First posted 2011-04-15 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-07

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome; Respiratory Failure
Keywords: Acute Lung Injury; Acute Respiratory Distress Syndrome; Respiratory Failure; Cytomegalovirus seropositive; Infection; Intravenous Ganciclovir; Non-immunocompromised; Valganciclovir
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Respiratory Insufficiency; Infections | interventions — Ganciclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV Ganciclovir (Experimental): 5mg/kg IV twice daily for 5 days, then followed by either IV ganciclovir or oral valganciclovir once daily until hospital discharge
  Interventions: Drug: IV Ganciclovir
- Placebo (Placebo Comparator): normal saline IV twice daily for 5 days, then followed by either IV normal saline or oral placebo once daily until hospital discharge
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IV Ganciclovir — For first 5 days, dosing of intravenous ganciclovir is 10 mg/kg daily, given as 5 mg/kg every 12 hours (adjusted for renal function). After first 5 days (up to 28 days) IV ganciclovir 5 mg/kg QD ( adjusted for renal function). A minimum interval of 6 hours is required between the first and second dose.
  Arms: IV Ganciclovir
Drug: Placebo — For first 5 days, dosing of intravenous placebo is daily, given every 12 hours. After first 5 days (up to 28 days), IV placebo QD. A minimum interval of 6 hours is required between the first and second dose.
  The placebo is an IV solution that does not contain any active medications.
  Arms: Placebo

SUMMARY:
To evaluate whether administration of ganciclovir reduces serum IL-6 levels (i.e. reduction between baseline and 14 days post-randomization) in immunocompetent adults with severe sepsis or trauma associated respiratory failure.

Primary Hypotheses:

- In CMV seropositive adults with severe sepsis or trauma , pulmonary and systemic CMV reactivation amplifies and perpetuates both lung and systemic inflammation mediated through specific cytokines, and contributes to pulmonary injury and multiorgan system failure,

AND

- Prevention of CMV reactivation with ganciclovir decreases pulmonary and systemic inflammatory cytokines that are important in the pathogenesis of sepsis and trauma related complications.

DETAILED DESCRIPTION:
Critical illness due to severe sepsis and trauma are major causes of morbidity and mortality, and a substantial economic burden in the United States and worldwide. Despite advances in clinical care, patients with sepsis and trauma-associated respiratory failure represent specific populations with high rates of adverse outcomes. The etiology of respiratory failure in patients with severe sepsis and trauma is multifactorial, but acute lung injury (ALI) is one of the leading causes, and is associated with prolonged ICU and hospital stays, mortality, and long-term sequelae. Other than general supportive care, few specific interventions other than lung protective ventilation have been shown to improve outcomes in such patients. New approaches for understanding the pathogenesis and developing better therapies are urgently needed.

Acute Lung Injury (ALI) is a syndrome consisting of acute hypoxemic respiratory failure with bilateral pulmonary infiltrates that is associated with both pulmonary and nonpulmonary risk factors (eg. sepsis, trauma) and that is not due primarily to left atrial hypertension. Although a distinction between ALI and a more severe subtype (termed acute respiratory distress syndrome (ARDS) has been made, the pathogenesis, risk factors, and outcomes appear to be similar and for the purposes of this protocol, the term acute lung injury [ALI] will be used to encompass both entities. Accepted consensus definitions of ALI have been introduced and are now widely used for laboratory and clinical investigations of ALI. Acute Lung Injury (ALI) is defined as:

* PaO2/FiO2 <300
* Bilateral pulmonary infiltrates on chest x-ray
* Pulmonary Capillary Wedge Pressure <18mmHg or no clinical evidence of increased left atrial pressure Although a broad range of risk factors for ALI have been described, those that account for the majority of cases include: sepsis, pneumonia, trauma, and aspiration. It is well established that severe trauma is recognized as a precipitating cause of ALI. Recent studies have demonstrated that the incidence of acute lung injury (ALI) is much higher than previously thought, with an estimated age-adjusted incidence of 86 per 100,000 persons per year, resulting in an estimated ~190,000 cases annually in the US. The clinical and health care system impact of ALI is substantial, with an estimated 2,154,000 intensive care unit (ICU) days, 3,622,000 hospital days, and 75,000 deaths in 2000, and is expected to grow significantly given the marked age-related incidence and the aging population. Although general improvements in ICU care over the last 2 decades have led to a trend towards lower mortality due to certain ALI-associated risk factors (trauma, aspiration), the most common causes of ALI, sepsis and pneumonia, remain associated with high mortality rates of ~25-35%. Mortality in ALI is most commonly due to secondary infections/sepsis and multiorgan system failure rather than primary respiratory failure due to hypoxemia, highlighting the systemic nature of ALI. Even among initial survivors of ALI, substantial pulmonary and nonpulmonary functional impairment remains for months to years. Specifically, a proportion of those who survive the initial insult are at risk for prolonged mechanical ventilation and ICU/hospital stay, and the risk factors remain poorly defined. It has been hypothesized that a "2nd hit" may predispose certain patients to greater morbidity in this setting. Despite intensive basic and clinical investigation, only a single intervention (low-tidal volume ["lung protective"] ventilation) is generally accepted to decrease mortality in ALI, while multiple other strategies have failed to improve survival either in early clinical studies or definitive efficacy trials. Thus, given the high incidence and continued substantial clinical impact of ALI despite improvements in general medical/ICU care, and limited proven options other than lung-protective ventilation, new approaches to understanding the pathophysiology and identifying novel targets for intervention in ALI are a high priority.

Overly intense, persistent and dysregulated pulmonary and systemic inflammation has emerged as the leading hypothesis for the pathogenesis of ALI and its complications, but the contributory factors and mechanisms are incompletely defined. Several carefully-conducted prospective human studies have shown an association between specific inflammatory biomarkers in blood and BALF (both the initial levels at onset and changes over time) and important clinical outcomes in ALI. [Animal models have also demonstrated an association between inflammatory cytokines and non-pulmonary organ injury and dysfunction] In addition, one of the most important interventions (low-tidal volume ["lung protective"] ventilation) shown to decrease mortality in ALI is associated with reductions in inflammatory cytokines (IL-6, IL-8) in blood and bronchoalveolar lavage fluid [BALF].

Cytomegalovirus (CMV) is a ubiquitous virus in humans worldwide, and has been linked to adverse clinical outcomes including prolongation of mechanical ventilation, increased length of stay, and mortality in multiple studies of critically-ill, apparently immunocompetent, seropositive adults.

Cytomegalovirus (CMV) is a human herpes virus known to infect more than 50-90% of US adults and is known to be a major cause of morbidity and mortality in immunocompromised patients. CMV infection can be acquired through multiple means, including: mother-to-child (in utero, breast milk), infected body fluids (saliva, genital secretions), blood transfusion or organ transplant. The prevalence of CMV infection increases with age throughout life such that by age 90, ~90% of persons will have acquired CMV infection. In immunocompetent persons, following primary infection by any of the routes noted above, CMV is controlled by the immune system and establishes latency ("dormancy") in multiple organs/cell-types for the life of the host. In particular, the lung represents one of the largest reservoirs of latent CMV in seropositive hosts, and may explain the propensity for CMV-associated pulmonary disease in predisposed hosts. During periods of immunosuppression (or as a result of specific stimuli such as TNF-α, LPS, or catecholamines that are commonly associated with critical illness & sepsis [CMV can reactivate from latency (preferentially in the lung) to produce active infection (viral replication). In persons with impaired cellular immunity, reactivation can progress to high-grade CMV replication and commonly leads to tissue injury and clinically-evident disease such as CMV pneumonia. Lower-grade CMV reactivation that is otherwise clinically silent ("subclinical") can also be detected in apparently immunocompetent persons with critical illness using sensitive techniques such as PCR. In addition, even low-level, otherwise asymptomatic subclinical CMV reactivation can produce significant biologic effects both in vitro and in vivo, such as inflammation, fibrosis and immunosuppression. Each of these biologic effects of subclinical CMV infection has either previously been demonstrated (inflammation, fibrosis) or could theoretically be important (immunosuppression) in sepsis-associated ALI and its complications. These biological effects of CMV have been shown to occur through various mediators and other indirect means [Importantly, several important CMV-associated adverse clinical outcomes in transplant populations [allograft rejection, secondary infections] are not necessarily accompanied by overt CMV disease and can only be detected by relatively sensitive means of virus detection such as PCR.

Reactivation of CMV in apparently immunocompetent patients with critical illness due to a broad range of causes has been documented in multiple prior studies using a variety of virologic techniques. The specific triggers for CMV reactivation from latency have been identified and are known to be elevated in patients with sepsis and acute lung injury [A prospective study in intubated patients with sepsis from Germany reported more than 60% rate of CMV DNA detection in tracheal aspirates.

In addition to CMV reactivation in sepsis, CMV reactivation has also been demonstrated specifically in lung and blood of patients with acute lung injury.

Retrospectively testing samples collected in a prospective observational cohort study of patients at risk of developing ARDS, CMV reactivation (ie. CMV DNA by PCR) was detected in BALF and/or plasma of 2/5 [40%] of subjects who developed ARDS, in sequential samples from 7/20 [35%] patients with ARDS, but not in patients at risk but who did not develop ARDS (0/5) [Limaye 2009 unpublished data]. In a separate study, CMV reactivation was retrospectively assessed by PCR in BALF of 88 subjects enrolled in a randomized trial of fish oil for treatment of ALI. Seropositivity at baseline (ie. evidence of latent CMV infection) in the cohort was 65% (similar to prior age-related estimates), and CMV reactivation (ie. CMV DNA by PCR) was detected in BALF of 12/57 [21%] patients [Limaye unpublished data 2009].

Several lines of evidence have linked CMV reactivation with adverse clinical outcomes in non-immunosuppressed adults with critical illness. In a recent meta-analysis, CMV reactivation (compared to no reactivation) was associated with a 2-fold increased odds of mortality in ICU patients.

In addition to mortality, recent studies have demonstrated a strong and independent association between CMV reactivation and increased hospital and ICU length of stay and duration of mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject/next of kin informed consent
2. Age >= 18 years
3. CMV IgG seropositive. The following tests are acceptable:

   * FDA licensed test in a local lab approved by the coordinating center (FHCRC, Seattle, WA).
   * Test in central study lab (ARUP, Salt Lake City, UT)
   * A report that patient has previously been tested and found to be CMV seropositive at any time (a credible next of kin report is acceptable; confirmatory test will be done but results are not required for randomization)
4. Intubated and requiring mechanical positive pressure ventilation (including Acute Lung Injury/ARDS (EA Consensus Definition))
5. Meets criteria for either:

   1. Severe sepsis criteria (as defined in appendix G) within a 24-hour time period within the 120 hour window

      OR
   2. Trauma with respiratory failure and an ISS score > 15 within a 24 hour time period, and within the 120 hour window (where mechanical ventilation is not due solely to a head injury)
6. On the day of randomization (by local criteria):

   * Not eligible for SBT (use of sedation and/or vasopressor does not specifically contraindicate SBT),or
   * Failed SBT

Exclusion Criteria:

1. BMI > 60 (1st weight during hospital admission)
2. Known or suspected immunosuppression, including:

   * HIV+ (i.e. prior positive test or clinical signs of suspicion of HIV/AIDS; a negative HIV test is not required for enrollment)
   * stem cell transplantation:

     * within 6 months after autologous transplantation or
     * within 1 years after allogeneic transplantation (regardless of immunosuppression)
     * greater than 1 year of allogeneic transplantation if still taking systemic immunosuppression or prophylactic antibiotics (e.g. for chronic graft versus host disease)

   Note: if details of stem cell transplantation are unknown, patients who do not take systemic immunosuppression and do not take anti-infective prophylaxis are acceptable for enrollment and randomization.
   * solid organ transplantation with receipt of systemic immunosuppression (any time).
   * cytotoxic anti-cancer chemotherapy within the past three months (Note: next-of-kin estimate is acceptable).
   * congenital immunodeficiency requiring antimicrobial prophylaxis (e.g. TMP-SMX, dapsone, antifungal drugs, intravenous immunoglobulin).
   * receipt of one or more of the following in the indicated time period:

     * within 6 months: alemtuzumab, antithymocyte/antilymphocyte antibodies
     * within 3 months: immunomodulator therapy (TNF-alpha antagonist, rituximab, tocilizumab, IL1 receptor antagonist and other biologics)
     * within 30 days:

       * corticosteroids > 10 mg/day (chronic administration, daily average over the time period)

         * topical steroids are permissible
         * use of hydrocortisone in "stress doses" up to 100 mg four times a day (400mg/daily) for up to 4 days prior to randomization is permissible
         * use of temporary short-term (up to 2 weeks) increased doses of systemic steroids (up tp 1 mg/kg) for exacerbation of chronic conditions are permissible.
       * methotrexate (> 10.0 mg/week)
       * azathioprine (> 75 mg/day)

   Note: if no information on these agents is available in the history and no direct or indirect evidence exists from the history that any condition exists that requires treatment with these agents (based on the investigator's assessment), the subject may be enrolled. For all drug information, next-of-kin estimates are acceptable. See Appendix D for commonly prescribed immunosuppressive agents.
3. Expected to survive < 72 hours (in the opinion of the investigator)
4. Has been hospitalized for > 120 hours (subjects who are transferred from a chronic care ward, such as a rehabilitation unit, with an acute event are acceptable).
5. Pregnant or breastfeeding (either currently or expected within one month).

   Note: for women of childbearing age (18-60 years, unless documentation of surgical sterilization [hysterectomy, tubal ligation, oophorectomy]), if a pregnancy test has not been done as part of initial ICU admission work-up, it will be ordered stat and documented to be negative before randomization. Both urine and blood tests are acceptable.
6. Absolute neutrophil count < 1,000/mm3 (if no ANC value is available, the WBC must be > 2500/mm3)
7. Use of cidofovir within seven (7) days of patient randomization. The use of the following antivirals is permitted under the following conditions:

   * Ganciclovir, foscarnet, high-dose acyclovir, or valacyclovir until the day of randomization
   * Acyclovir as empiric therapy for central nervous system HSV or VZV infection until the diagnosis can be excluded
   * For enrolled patients during the active study drug phase, acyclovir, famciclovir, valacyclovir for treatment of HSV or VZV infection as clinically indicated.
8. Currently enrolled in an interventional trial of an investigational therapeutic agent known or suspected to have anti-CMV activity, or to be associated with significant known hematologic toxicity (Note: confirm eligibility with one of the study medical directors at the coordinating site).
9. At baseline patients who have both a tracheostomy, and have been on continuous 24-hour chronic mechanical ventilation.
10. Patients with Child Class C Cirrhosis.
11. Patients with pre-existing interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-03-10 (Actual); Primary Completion 2016-06-17 (Actual); Study Completion 2016-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boeckh, MD, Principal Investigator — Fred Hutchinson Cancer Center; Ajit Limaye, MD, Principal Investigator — University of Washington; Louise Kimball, PhD, RN, Study Director — Fred Hutchinson Cancer Center
Locations (14):
- United States (14):
  - University of Colorado / National Jewish Health / Swedish Medical Center, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - Baystate Critical Care Medicine / Tufts University School of Medicine, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Wakeforest University, School of Medicine, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - The Oregon Clinic, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Vermont College of Medicine, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Harborview Medical Center, Seattle, Washington
  - University of Washington Medical Center / Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Limaye AP, Stapleton RD, Peng L, Gunn SR, Kimball LE, Hyzy R, Exline MC, Files DC, Morris PE, Frankel SK, Mikkelsen ME, Hite D, Enfield KB, Steingrub J, O'Brien J, Parsons PE, Cuschieri J, Wunderink RG, Hotchkin DL, Chen YQ, Rubenfeld GD, Boeckh M. Effect of Ganciclovir on IL-6 Levels Among Cytomegalovirus-Seropositive Adults With Critical Illness: A Randomized Clinical Trial. JAMA. 2017 Aug 22;318(8):731-740. doi: 10.1001/jama.2017.10569. PMID 28829877

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: normal saline IV twice daily for 5 days, then followed by either IV normal saline or oral placebo once daily until hospital discharge
  Placebo: For first 5 days, dosing of intravenous placebo is daily, given every 12 hours. After first 5 days (up to 28 days), IV placebo QD. A minimum interval of 6 hours is required between the first and second dose.
  The placebo is an IV solution that does not contain any active medications.
Period: Overall Study
Arm/Group | IV Ganciclovir | Placebo
Started | 84 | 76
Completed | 84 | 72
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Ganciclovir | Placebo | Total
Number analyzed (Participants) | 84 | 76 | 160
Age, Continuous [Mean (Full Range); unit: years] | 55.2 [18 to 95] | 58.2 [18 to 95] | 56.6 [18 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 71
  Male | 49 | 40 | 89
Region of Enrollment [Number; unit: participants]
  United States | 84 | 76 | 160

OUTCOME MEASURES:

1. Primary Outcome: Serum IL-6 Level
Description: Change between baseline and 14 days post-randomization between placebo & ganciclovir groups
Time Frame: Baseline and Day 14
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
pg/mL | -0.79 (0.65) | -0.79 (0.69)

2. Secondary Outcome: Number of Participants With CMV Reactivation at 28 Days in Plasma
Description: Number of participants in baseline negatives with CMV reactivation at any level at day 28
Time Frame: at 28 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 77 | 67
Participants
  CMV viremia at any level | 3 | 23
  no CMV viremia at any level | 74 | 44
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = .0001, Fisher Exact

3. Secondary Outcome: BAL Levels of IL-6
Description: Levels of IL-6 from BALs at 7 days post-randomization
Time Frame: at 7 days post-randomization
Population: The protocol was modified to remove the inclusion of BALs, thus these numbers reflect the total BALs performed prior to the modification.
Measure: Mean (Standard Deviation); unit: log 10 pg/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 3 | 7
log 10 pg/mL | 1.01 (0.78) | 1.66 (1.26)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.31, t-test, 2 sided

4. Secondary Outcome: Number of Participants With Organ System Failure at 14 Days
Description: Number of participants experiencing organ system failure at 14 days
Time Frame: at 14 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
Participants
  with organ failure | 0 | 2
  without organ failure | 84 | 70

5. Secondary Outcome: Number of Days Alive and Not in the ICU
Description: Number of ICU days alive and not in the ICU by day 28
Time Frame: by 28 days post-randomization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
days | 10.02 (6.84) | 10.97 (8.23)

6. Secondary Outcome: CMV Disease
Description: Need to be biopsy-proven
Time Frame: by 180 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
Participants
  Biopsy proven CMV disease | 0 | 0
  No Biopsy proven CMV disease | 84 | 72

7. Secondary Outcome: Grade 3 AEs or Higher
Description: Number of patients with greater than one AE of grade 3 or more
Time Frame: by 35 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
Participants
  number with AE greater than grade 3 | 11 | 10
  number without AE greater than grade 3 | 73 | 62

8. Secondary Outcome: SF-36 Health Survey
Description: Physical Component Summary of SF-36. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Time Frame: at 1 day post-randomization
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 53 | 35
scores on a scale | 36.37 (10.93) | 35 (11.28)

9. Secondary Outcome: Incidence of CMV Reactivation >1,000 IU Per mL at Day 28 in Plasma
Description: Number of participants with CMV reactivation >1,000 IU per mL at day 28 in plasma
Time Frame: at 28 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 77 | 67
Participants
  CMV viremia >1,000 copies per mL | 0 | 5
  No CMV viremia >1,000 copies per mL | 77 | 62
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.006, Fisher Exact

10. Secondary Outcome: Incidence of CMV Reactivation at Any Level at 28 Days in Throat
Description: CMV reactivation in baseline negatives at any level at day 28 in throat
Time Frame: at 28 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 80 | 67
Participants
  CMV reactivation at any level at day 28 in throat | 2 | 6
  No CMV reactivation at any level at day 28in throa | 78 | 61
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.14, Fisher Exact

11. Secondary Outcome: Incidence of CMV Reactivation >1,000 IU Per mL at 28 Days in Throat
Description: Number of participants with CMV reactivation >1,000 IU per mL at day 28 in throat
Time Frame: at 28 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 80 | 67
Participants
  CMV reactivation >1,000 in IU per mL | 0 | 1
  No CMV reactivation >1,000 IU per mL in throat | 80 | 66
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.10, Fisher Exact

12. Secondary Outcome: CMV AUC in Blood
Description: CMV AUC in blood from day 0 to day 28
Time Frame: Day 0 to 28 days post-randomization
Measure: Mean (Standard Deviation); unit: IU*day/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
IU*day/mL | 0.11 (0.39) | 0.39 (0.69)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.002, t-test, 2 sided

13. Secondary Outcome: CMV AUC in Throat
Description: CMV AUC in Throat from day 0 to day 28
Time Frame: Day 0 to 28 days post-randomization
Measure: Mean (Standard Deviation); unit: IU*day/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
IU*day/mL | 0.03 (0.14) | 0.17 (0.52)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.03, t-test, 2 sided

14. Secondary Outcome: CMV Peak Viral Load in Blood
Description: CMV Peak Viremia in blood at day 28
Time Frame: at 28 days post-randomization
Measure: Mean (Standard Deviation); unit: log 10 IU/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
log 10 IU/mL | 0.24 (0.67) | 0.89 (1.21)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p < 0.0001, t-test, 2 sided

15. Secondary Outcome: BAL Levels of IL-8
Description: Levels of IL-8 in BALs at day 7
Time Frame: at 7 days post-randomization
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log 10 pg/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 3 | 7
log 10 pg/mL | 2.21 (0.66) | 2.61 (1.22)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.73, t-test, 2 sided

16. Secondary Outcome: BAL Levels of TNFa
Description: Levels of TNFa in BALs at day 7
Time Frame: at 7 days post-randomization
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log 10 pg/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 3 | 7
log 10 pg/mL | 0.18 (0) | 0.46 (0.49)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.33, t-test, 2 sided

17. Secondary Outcome: Plasma Levels of IL-6
Description: Plasma levels of IL-6.
Time Frame: at 7 days post-randomization
Measure: Mean (Standard Deviation); unit: log 10 pg/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 75 | 57
log 10 pg/mL | 0.87 (0.84) | 0.92 (0.62)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.31, t-test, 2 sided

18. Secondary Outcome: Plasma Levels of IL-8
Description: Levels of IL-8 in plasma at day 7
Time Frame: at 7 days post-randomization
Measure: Mean (Standard Deviation); unit: log 10 pg/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 75 | 57
log 10 pg/mL | 1.38 (0.6) | 1.38 (0.35)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.96, t-test, 2 sided

19. Secondary Outcome: Plasma Levels of TNF a
Description: Plasma levels of TNF a at day 7.Cytokines are summarized on log 10 scale. When logged value is negative, the raw value would be less than 1.
Time Frame: at 7 days post-randomization
Measure: Mean (Standard Deviation); unit: log 10 pg/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 75 | 57
log 10 pg/mL | -0.07 (0.36) | -0.1 (0.35)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.63, t-test, 2 sided

20. Secondary Outcome: Plasma Levels of TNF a
Description: Plasma levels of TNF a from day 0 to day 28
Time Frame: Day 0 to 28 days post-randomization
Population: Cytokines are summarized on a log 10 scale. When the logged value is negative, the raw value would be less than 1.
Measure: Mean (Standard Deviation); unit: log 10 pg/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 33 | 31
log 10 pg/mL | -0.06 (0.37) | -0.11 (0.27)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.51, t-test, 2 sided

21. Secondary Outcome: Plasma Levels of IL-6
Description: Plasma levels of IL-6 at day 28
Time Frame: at 28 days post-randomization
Measure: Mean (Standard Deviation); unit: log 10 pg/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 33 | 31
log 10 pg/mL | 0.35 (0.51) | 0.59 (0.7)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.12, t-test, 2 sided

22. Secondary Outcome: Plasma Levels of IL-8
Description: Plasma levels of IL-8 at day 28
Time Frame: at 28 days post-randomization
Measure: Mean (Standard Deviation); unit: log 10 pg/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 33 | 31
log 10 pg/mL | 1.09 (0.46) | 1.27 (0.46)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.13, t-test, 2 sided

23. Secondary Outcome: Plasma Levels of Soluble ICAM-1
Description: Plasma levels of soluble ICAM-1 at day 28
Time Frame: at 28 days post-randomization
Measure: Mean (Standard Deviation); unit: log 10 pg/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 33 | 31
log 10 pg/mL | 5.34 (0.19) | 5.48 (0.22)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.008, t-test, 2 sided

24. Secondary Outcome: Plasma Levels of Soluble ICAM-1
Description: Plasma levels of soluble ICAM-1 at day 7
Time Frame: at 7 days post-randomization
Measure: Mean (Standard Deviation); unit: log 10 pg/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 75 | 57
log 10 pg/mL | 5.43 (0.21) | 5.45 (0.31)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.64, t-test, 2 sided

25. Secondary Outcome: Peak Plasma Levels of Soluble ICAM-1
Description: Peak Plasma levels of soluble ICAM-1 from day 0 to day 28
Time Frame: Day 0 to 28 days post-randomization
Measure: Mean (Standard Deviation); unit: log 10 pg/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
log 10 pg/mL | 5.52 (0.2) | 5.57 (0.27)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.24, t-test, 2 sided

26. Secondary Outcome: Peak Plasma Levels of TNF-a
Description: Peak Plasma levels of TNF-a at day 28
Time Frame: at 28 days post-randomization
Measure: Mean (Standard Deviation); unit: log 10 pg/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
log 10 pg/mL | 0.16 (0.3) | 0.17 (0.36)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.76, t-test, 2 sided

27. Secondary Outcome: Peak Plasma Levels of IL-10
Description: Peak Plasma levels of IL-10 at day 28
Time Frame: at 28 days post-randomization
Measure: Mean (Standard Deviation); unit: log 10 pg/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
log 10 pg/mL | 0.88 (0.52) | 0.82 (0.49)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.45, t-test, 2 sided

28. Secondary Outcome: Peak Plasma Levels of IL-8
Description: Peak Plasma levels of IL-8 at day 28
Time Frame: at 28 days post-randomization
Measure: Mean (Standard Deviation); unit: log 10 pg/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
log 10 pg/mL | 1.67 (0.65) | 1.66 (0.44)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.92, t-test, 2 sided

29. Secondary Outcome: Peak Plasma Levels of IL-6
Description: Peak Plasma levels of IL-6 at day 28
Time Frame: at 28 days post-randomization
Measure: Mean (Standard Deviation); unit: log 10 pg/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
log 10 pg/mL | 1.57 (0.78) | 1.56 (0.78)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.94, t-test, 2 sided

30. Secondary Outcome: AUC Plasma Levels of IL-6
Description: AUC Plasma levels of IL-6 from day 0 to day 28
Time Frame: Day 0 to 28 days post-randomization
Measure: Mean (Standard Deviation); unit: IU*day/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
IU*day/mL | 0.68 (0.49) | 0.75 (0.51)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.37, t-test, 2 sided

31. Secondary Outcome: AUC Plasma Levels of IL-8
Description: AUC Plasma levels of IL-8 from day 0 to day 28
Time Frame: Day 0 to 28 days post-randomization
Measure: Mean (Standard Deviation); unit: IU*day/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
IU*day/mL | 1.15 (0.45) | 1.13 (0.42)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.80, t-test, 2 sided

32. Secondary Outcome: AUC Plasma Levels of IL-10
Description: AUC Plasma levels of IL-10 from day 0 to day 28
Time Frame: at 28 days post-randomization
Measure: Mean (Standard Deviation); unit: IU*day/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
IU*day/mL | 0.36 (0.36) | 0.35 (0.38)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.93, t-test, 2 sided

33. Secondary Outcome: AUC Plasma Levels of TNF-a
Description: AUC Plasma levels of TNF-a from day 0 to day 28
Time Frame: at 28 days post-randomization
Measure: Mean (Standard Deviation); unit: IU*day/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
IU*day/mL | -0.14 (0.28) | -0.14 (0.25)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.93, t-test, 2 sided

34. Secondary Outcome: AUC Plasma Levels of Soluble ICAM-1
Description: AUC Plasma levels of soluble ICAM-1 from day 0 to day 28
Time Frame: at 28 days post-randomization
Measure: Mean (Standard Deviation); unit: IU*day/mL
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
IU*day/mL | 4.78 (0.98) | 4.65 (1.25)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Other; p = 0.45, t-test, 2 sided

35. Secondary Outcome: Length of Stay
Description: Hospital days alive and not hospitalized by day 180
Time Frame: by 180 days post-randomization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 55 | 47
days | 145.13 (47.63) | 145.94 (47.88)

36. Secondary Outcome: Length of Stay
Description: Hospital days alive and not hospitalized by day 28
Time Frame: by 28 days post-randomization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 78 | 69
days | 9.96 (8.52) | 8.72 (8.24)

37. Secondary Outcome: Organ System Failure at 28 Days
Description: Number of participants with organ system failure at 28 days
Time Frame: at 28 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
Participants
  with organ failure | 0 | 2
  without organ failure | 84 | 70

38. Secondary Outcome: Duration of Mechanical Ventilation as Assessed by Ventilator Free Days
Description: Number of days of mechanical ventilation duration as assessed by ventilator free days
Time Frame: at 28 days post-randomization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
days | 18.71 (9.08) | 15.97 (9.72)

39. Secondary Outcome: Duration of Mechanical Ventilation as Assessed by Ventilator Days
Description: Number of days of mechanical ventilation duration as assessed by ventilator days
Time Frame: at 28 days post-randomization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
days | 6.95 (6.16) | 8.5 (7.17)

40. Secondary Outcome: Bacteremia and/or Fungemia
Description: Number of participants with bacteremia and/or fungemia
Time Frame: at 28 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
Participants
  with bacteremia and /or fungemia | 15 | 11
  without bacteremia and /or fungemia | 69 | 61

41. Secondary Outcome: Mortality
Description: Mortality at 60 days post randomization
Time Frame: at 60 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
Participants
  dead | 13 | 12
  alive | 71 | 60

42. Secondary Outcome: Mortality at 180 Days
Description: Mortality at 180 days post-randomization
Time Frame: at 180 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
Participants
  dead | 18 | 19
  alive | 66 | 53

43. Secondary Outcome: SF-36 Functional Assessment Physical Component
Description: Physical Component Summary at 180 days post- randomization. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability
Time Frame: at 180 days post-randomization
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 40 | 34
scores on a scale | 35.51 (11.38) | 38.17 (10.96)

44. Secondary Outcome: SF-36 Functional Assessment Mental Component
Description: Mental Component Summary at 180 days post-randomization. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability
Time Frame: at 180 days post-randomization
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 40 | 34
scores on a scale | 45.55 (11.52) | 44.08 (12.25)

45. Secondary Outcome: SF-36 Functional Assessment Mental Component on Day 1
Description: SF-36 Mental Component Summary at 1 day post-randomization. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability
Time Frame: at 1 day post-randomization
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 53 | 35
scores on a scale | 43.83 (12) | 42.73 (13.78)

46. Secondary Outcome: Patients With Serious Adverse Events
Description: Number of patients with Serious Adverse Events by day 35
Time Frame: by 35 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
Participants
  Number of patients with a Serious adverse event | 0 | 0
  Number of patients without a Serious adverse event | 84 | 72

47. Secondary Outcome: Time to Neutropenia
Description: Time to neutropenia by 35 days post-randomization
Time Frame: by 35 days post-randomization
Measure: Number; unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
days | 0 | 0

48. Secondary Outcome: Use of Granulocyte-colony Stimulating Factor
Description: Number of participants requiring Granulocyte-colony stimulating factor
Time Frame: by 35 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
Participants
  Number of patients that required GCSF | 0 | 0
  Number of patients that did not require GCSF | 84 | 72

49. Secondary Outcome: Renal Insufficiency
Description: Number of patients experiencing a glomerular filtration rate < 60mL/min at day 35
Time Frame: by 35 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
Participants
  Glomerular filtration rate less than 60 mL/min | 36 | 41
  Glomerular filtration rate greater than 60 mL/min | 48 | 31

50. Secondary Outcome: Red Blood Cell Transfusions Required Per Patients
Description: Red blood cell transfusions required per patients by day 35
Time Frame: by 35 days post-randomization
Measure: Median (Inter-Quartile Range); unit: transfusions
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
transfusions | 2 [1 to 2] | 1 [1 to 4]

51. Secondary Outcome: Platelet Transfusions
Description: Platelet transfusions per patient
Time Frame: by 35 days post-randomization
Measure: Median (Inter-Quartile Range); unit: transfusions
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 721
transfusions | 1 [1 to 1] | 1 [1 to 2]

52. Secondary Outcome: Clinical Outcomes
Description: Composite of survival status and >7 days ventilation status, and IL-6 levels. In the composite analysis, the endpoint is composed by death, ventilation status and change of cytokine.
Time Frame: at 14 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 84 | 72
Participants
  Number of patients with composite endpoint | 42 | 49
  Number of patients without composite endpoint | 42 | 23

53. Secondary Outcome: Bacteremia and Fungemia Outcomes
Description: Bacteremia and fungemia outcomes among subjects who survive at least 7 days
Time Frame: at 7 days post-randomization
Measure: Number; unit: events
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 82 | 64
events
  number of events | 15 | 9
  number of no events | 67 | 55

54. Secondary Outcome: Bacteremia and Fungemia Outcomes in Mechanically Ventilated Subjets
Description: Bacteremia and fungemia events among subjects who are mechanically ventilated for at least 7 through 14 days after randomization
Time Frame: at 7 through 14 days post-randomization
Measure: Number; unit: events
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 30 | 33
events
  number of events | 6 | 9
  number of no events | 24 | 24

55. Secondary Outcome: Overall Mortality
Description: Overall mortality amongst subjects who survive at least 7 days after randomization
Time Frame: at 7 days post-randomization
Measure: Number; unit: events
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 82 | 64
events
  number of deaths | 16 | 11
  number of alive | 66 | 53

56. Secondary Outcome: Number of Mechanical Ventilated Days
Description: Number of mechanical ventilated days amongst subjects who survive at least 7 days after randomization
Time Frame: at 7 days post-randomization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 82 | 64
days | 7.05 (6.19) | 9.05 (7.4)

57. Secondary Outcome: Number of Ventilator-free Days
Description: Number of ventilator-free days amongst subjects who survive at least 7 days after randomization
Time Frame: at 7 days post-randomization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 82 | 64
days | 19.17 (8.7) | 17.97 (8.37)

58. Secondary Outcome: Number of Days in the ICU
Description: Number of days in the ICU amongst subjects who survive at least 7 days after randomization
Time Frame: at 7 days post-randomization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 82 | 64
days | 10.20 (6.82) | 11.83 (8.32)

59. Secondary Outcome: Number of ICU-free Days
Description: Number of ICU-free days amongst subjects who survive at least 7 days after randomization
Time Frame: at 7 days post-randomization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 82 | 64
days | 15.38 (27) | 13.89 (25)

60. Secondary Outcome: Number of Days in the Hospital
Description: Number of days in the hospital amongst subjects who survive at least 7 days after randomization
Time Frame: at 7 days post-randomization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 67 | 57
days | 6.21 (4.85) | 5.53 (4.9)

61. Secondary Outcome: Number of Hospital-free Days
Description: Number of hospital-free days amongst subjects who survive at least 7 days after randomization
Time Frame: at 7 days post-randomization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 76 | 61
days | 10.22 (8.47) | 9.87 (8.09)

62. Secondary Outcome: Mortality Among Subjects Mechanically Ventilated From Day 7 to 14
Description: Mortality among subjects by day 28 who are mechanically ventilated for at least 7 through 14 days after randomization
Time Frame: 28 days
Measure: Number; unit: events
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 30 | 33
events
  number of events | 9 | 6
  number of no events | 21 | 27

63. Secondary Outcome: Number of Mechanically Ventilated Days Among Subjects by Day 28
Description: Number of mechanically ventilated days among subjects by day 28 who are mechanically ventilated for at least 7 through 14 days after randomization
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 30 | 33
days | 13.4 (6.12) | 14.42 (6.64)

64. Secondary Outcome: Number of Ventilator-free Days Among Subjects by Day 28
Description: Number of ventilator-free days among subjects by day 28 who are mechanically ventilated for at least 7 through 14 days after randomization
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 30 | 33
days | 11.4 (8.29) | 12.45 (7.26)

65. Secondary Outcome: Number of Days in ICU Amongst Subjects by Day 28
Description: Number of days in ICU amongst subjects by day 28 who are mechanically ventilated for at least 7 through 14 days after randomization
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 30 | 33
days | 16.73 (5.75) | 17.79 (7.41)

66. Secondary Outcome: Number of ICU-free Days Amongst Subjects by Day 28
Description: Number of ICU-free days amongst subjects by day 28 who are mechanically ventilated for at least 7 through 14 days after randomization
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 30 | 33
days | 7.73 (18) | 8.15 (18)

67. Secondary Outcome: Number of Hospital-free Days Among Subjects by Day 28
Description: Number of hospital-free days among subjects by day 28 who are mechanically ventilated for at least 7 through 14 days after randomization
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 28 | 32
days | 3.54 (5.15) | 4.59 (5.55)

ADVERSE EVENTS:
Time Frame: Clinical adverse events were collected from day 1(start of study drug) through day 35 (7 days after the stop of study drug).
Arm/Group | IV Ganciclovir | Placebo
All-Cause Mortality (participants affected / at risk) | 10/84 | 11/72
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/72
Other Adverse Events (participants affected / at risk) | 0/84 | 0/72

LIMITATIONS AND CAVEATS:
Inclusion of too few trauma patients to assess treatment effects, a long enrollment window length, discontinuation of BAL sampling due to feasibility and changes in oral drug availability (later part of the study)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No